CLINICAL TRIAL: NCT00872053
Title: Effect of Robot-assisted Training on Foot Drop in Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B4125K-1
Record Dates: First submitted 2009-03-27; First posted 2009-03-31 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: MS (Multiple Sclerosis)
Keywords: robot; treadmill; foot drop; rehabilitation; gait
MeSH Terms: conditions — Multiple Sclerosis; Peroneal Neuropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Focused Ankle Training
  Interventions: Device: Anklebot
- Arm 2 (Experimental): Combination Therapy
  Interventions: Device: Anklebot; Device: Lokomat

INTERVENTIONS:
Device: Anklebot — The Anklebot is a robotic device that is worn via a leather boot and knee brace (Fig.1). As the participant goes through a series of ankle-training "games," the Anklebot can assist ankle movement throughout 3 planes.
Device: Lokomat — The Lokomat is a motor driven exoskeleton device that employs a body weight support suspension system and treadmill. Attached to the lower limbs, the Lokomat moves the subject's legs over a treadmill through position controlled trajectories that mimic normal human gait patterns.
  Arms: Arm 2

SUMMARY:
The primary aim of this study is to:

1. Collect pilot data on the effect of task-specific lower extremity training using the Anklebot on subjects with Multiple Sclerosis (MS) and who have foot drop;
2. Collect pilot data on the use of combination therapy on improving gait in subjects with MS. This therapy will use both Anklebot training and robot-assisted gait training.

Hypothesis: Both trainings will result in improved walking performance, but the combination therapy will result in greater gains than ankle training alone.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MS by McDonald criteria (McDonald, Compston et al. 2001). EDSS level between 3.5-5.5, who report ambulation problems.
* Presence of unilateral foot drop that is clinically apparent to the PI or PI designate.
* Must be able to ambulate 25 feet without an assisting device.

Exclusion Criteria:

* Cardiovascular: recent MI < 4 wk, uncontrolled HTN >190/110 mmHg.
* History of uncontrolled diabetes.
* Symptoms of orthostasis when standing up.
* Circulatory problems, history of vascular claudication or pitting edema.
* Unable to fully understand instructions in order to use the equipment or the process of the study.
* Body weight over 150 kg.
* Lower extremity injuries that limit range of motion or function.
* Joint problems (hip or leg) that limit range of motion or cause pain with movement despite treatment.
* Unstable fractures.
* Pressure sores with any skin breakdown in areas in contact with the body harness or Lokomat apparatus.
* Chronic and ongoing alcohol or drug abuse.
* Pre-morbid, ongoing depression or psychosis.
* Ongoing physical therapy.
* Pregnancy (self-reported)
* PI's determination of inability to complete the test protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Ankle accuracy and stiffness | At inclusion, after 8 sessions, after 16 sessions

SECONDARY OUTCOMES:
Gait assessments (e.g., 6-Minute Walk, Timed 25-Foot Walk) | At inclusion, after every 4 sessions
Functional assessments (EDSS, MS Functional Composite) | At inclusion, after 8 sessions, after 16 sessions

CONTACTS AND LOCATIONS:
Overall Officials: Albert Lo, MD PhD, Principal Investigator — Providence VA Medical Center
Locations (1):
- Providence VA Medical Center, Providence, Rhode Island, United States